CLINICAL TRIAL: NCT00347737
Title: The Effects of Therapy With Teriparatide (Recombinant Parathyroid Hormone (1-34) on Vascular Compliance and Osteoprotegerin/RANKL
Brief Title: The Effects of Therapy With Teriparatide on Vascular Compliance and Osteoprotegerin/RANKL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Leland Graves III, MD (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor-Investigator, Leland Graves III, MD, Associate Professor and Division Director, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10386
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Teriparatide
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — Teriparatide
  Other Names: Forteo

SUMMARY:
The purpose of this study is to determine what effect teriparatide will have on vascular (blood vessel) compliance and osteoprotegerin (bone fluid)and RANKL levels (bone cells).

DETAILED DESCRIPTION:
Research subjects participation is about 6 months. Subjects will give themselves daily injections of teriparatide after instruction on technique.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women and men over the age of 40 who are starting therapy with teriparatide

Exclusion Criteria:

* Patients with diabetes mellitus
* current smokers
* patients with a history of organ transplantation
* Patients currently of previously on glucocorticoid therapy within the past year
* Patients with serum creatinine above 1.5 mg/dl, patients with uncontrolled hypertension (BP 140/90 or greater)
* Patients ineligible for teriparatide therapy: History of metabolic bone disease other than osteoporosis
* History of radiation therapy
* Patients pregnant or nursing
* History of bone metastasis or skeletal malignancies
* History of hypercalcemia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The study measures changes in vascular compliance with teriparatide 1 hour, 3 months, and 6 months after initiating teriparatide. Osteoprotegerin and RANKL levels | baseline, 3, and 6 months

SECONDARY OUTCOMES:
CRP levels | Baseline and at 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Leland Graves, III, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States